CLINICAL TRIAL: NCT04141982
Title: Clinical Concordance Evaluation of the T-SPOT®.TB Assay Performance Using Positive Selection With the T-Cell SelectTM Kit and Density Gradient Cell Isolation Methods
Brief Title: Clinical Concordance Evaluation of T-SPOT®.TB Assay Performance (T-Cell SelectTM Study)
Status: Completed | Type: Observational
Sponsor: Oxford Immunotec (Industry)
Responsible Party: Sponsor
Other Study IDs: OI-18-01-IP-0001
Record Dates: First submitted 2019-10-25; First posted 2019-10-28 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Suspected of having TB infection: These donors are suspected of having TB infection and live in a high endemic area for TB infection
  Interventions: Diagnostic Test: T-Cell SelectTM Kit
- No (or minimal) TB risk factors: These donors must have no previous medical record of TB infection and live in low endemic area for TB infection
  Interventions: Diagnostic Test: T-Cell SelectTM Kit
- low/intermediate risk of TB infection population: These donors must live in an low/intermediate endemic area for TB infection
  Interventions: Diagnostic Test: T-Cell SelectTM Kit

INTERVENTIONS:
Diagnostic Test: T-Cell SelectTM Kit — The T-Cell Select kit is intended for the isolation of mononuclear immune cells from whole blood, using positive selection via a magnetic bead-based cell separation system, for use in the T-SPOT.TB assay.

SUMMARY:
The objective is to achieve 90% overall, positive and negative clinical concordance between results of the T-SPOT.TB assay, using cells isolated via density gradient centrifugation and positive selection using the T-Cell Select kit, between 0-55 hours following venepuncture

DETAILED DESCRIPTION:
In this study, clinical concordance between results of the T-SPOT.TB assay, using cells stored for 0-8 hours post venepuncture and isolated via density gradient separation and positive selection with magnetic bead isolation using the T-Cell SelectTM Kit will be assessed. Concordance between results of the T-SPOT.TB assay at 0-8 hours post venepuncture and using cells isolated with density gradient centrifugation and results obtained from cells isolated using the T-Cell Select Kit, following storage between 0-55 hours post venepuncture, will be assessed.

ELIGIBILITY:
Subjects presenting at sites enrolling "suspected of having TB infection" population Inclusion Criteria

* Be able to provide informed consent
* Be able to provide a minimum of 7 mL and maximum of 20 mL of whole blood.
* Have suspected TB infection.
* Be at least 18 years of age.
* Live in a high endemic area for TB infection

Exclusion Criteria

• Unable to meet inclusion criteria

Subjects presenting at sites enrolling "no (or minimal) TB risk factors" population Inclusion Criteria

* Be able to provide informed consent
* Be able to provide a minimum of 7 mL and maximum of 20 mL of whole blood.
* Have no suspicion TB infection.
* Be at least 18 years of age.
* Live in low endemic area for TB infection
* Have no previous medical record of TB infection

Exclusion Criteria

* Unable to meet inclusion criteria
* Current/previous TB diagnosis

Subjects presenting at sites enrolling "low/intermediate TB risk factors" population Inclusion Criteria

* Be able to provide a minimum of 7 mL and maximum of 20 mL of whole blood.
* Have no suspicion TB infection.
* Be at least 18 years of age.
* Live in an low/intermediate endemic area for TB infection Exclusion Criteria
* Unable to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This evaluation will collect blood samples from subjects suspected of having TB infection and, samples from a low risk control population with no (or minimal) TB risk factors. All subjects presenting at participating clinics will be eligible for enrolment into the study provided they meet the inclusion/exclusion criteria outlined in section 4. Based on previous experience and the medical profile of the patient attending each of clinics at the four study sites, it is expected that the sites will individually, and collectively, yield a range of positive and negative assay results required to assess the impact of the T-Cell Select kit on positive and negative agreements of the T-SPOT.TB test.
Sampling Method: Probability Sample
Enrollment: 680 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Achieving positive and negative clinical concordance between results of the T-SPOT.TB assay between 0-55hours after venipuncture | 1 year
  Achieving 90% overall, positive and negative clinical concordance between results of the T-SPOT.TB assay, using cells isolated via density gradient centrifugation and positive selection using the T-Cell Select kit, between 0-55 hours following venepuncture

CONTACTS AND LOCATIONS:
Overall Officials: Andre Trollip, PhD, Principal Investigator — Rapitrade; Blanca Restrepo, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Ehab Sorial, MD, Principal Investigator — NECCR Primacare Research, LLC; Shu-Hua Wang, MD, Principal Investigator — Ohio State University
Locations (4):
- United States (3):
  - NECCR Primacare Research, LLC, Fall River, Massachusetts
  - Ohio State University, Columbus, Ohio
  - University of Texas Health Science Center at Houston, School of Public Health in Brownsville, Brownsville, Texas
- Rapitrade, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No